CLINICAL TRIAL: NCT02662101
Title: Molecular Microbial Ecology as a Diagnostic Tool to Identify Mode of Action and New Targets for Oxidized Silver Wound Dressings
Brief Title: Impact of Oxidized Silver Wound Dressings on Wound Bacteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exciton Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Engage-453139_2013
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm, exsalt application (Experimental)
  Interventions: Device: Exsalt SD7, Exsalt T7 Wound Dressing

INTERVENTIONS:
Device: Exsalt SD7, Exsalt T7 Wound Dressing

SUMMARY:
Chronic non-healing wounds considerably impact quality of life in affected patients and are a substantial burden on the Canadian health care system. Microbes colonizing a chronic wound play an important role in impeding effective healing. Chronic wounds are colonized by polymicrobial communities and no single organism can be seen as causal. Only a small fraction of wound bacteria are cultured by diagnostic tests and studies have shown little agreement between culture and molecular based approaches, therefore an effective diagnostic for wound microbes is required. It is know that the composition of the microbial community associated with a wound changes as it heals although the causal relationship is somewhat unclear. Although not very effective in treating chronic non-healing wounds, antibiotics are often administered, contributing to concerns of antibiotic resistance. The wound dressings produced by Exciton Technologies Inc. (ETI) effectively aid in the healing process in chronic wounds through unknown mechanisms. ETI's wound dressings contain a combination of silver salts with three different valence, +1, +2 and +3 that have antimicrobial activity and are effective in reducing biofilm formation in vitro. However, it is not known how these silver salts impact microbial ecology of the wound and the role this plays in wound healing. The objectives of this research are to develop a new diagnostic tool based on molecular characterization of wound sites so as to predict how to best treat wounds and to identify new microbes to be targeted by ETI's technology. This project will utilize molecular microbial ecology for the assessment and evaluation of topical silver interventions, gaining insight into the management of chronic infection. Substantiating the microbiota-modifying effectiveness of silver wound dressings towards increasing clinician and patient understanding to improving clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed or verbal informed consent
2. >17 yrs and <70 yrs of age
3. have a chronic wound (defined as >6 weeks, non-healing), with or without clinical signs of infection.
4. requires visitation or admittance to the clinic and subsequent visits for dressing changes

Exclusion Criteria:

1. Systemic antibiotics within the last 2 weeks.
2. known skin sensitivity to any of the dressing components
3. Poor prognosis and who are unlikely to survive the trial period.
4. Participating in another concurrent trial.
5. Exhibiting any other medical condition, which, according to the investigator, justifies the subject's exclusion from the trial.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Observe microbes in the wound | 4 weeks
  The primary outcome variable will be the observations to changes in the composition of microbes after the application of the wound dressing.

SECONDARY OUTCOMES:
Observe wound progression | 4 weeks
  The second outcome variables will measure wound progression and healing as measured by a standard wound assessment protocol used in the clinic and recorded with pixelere software

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Kalan, PhD, Study Chair — Exciton Technologies

IPD SHARING:
Plan to Share IPD: No